CLINICAL TRIAL: NCT06192485
Title: Proactive and Reactive Balance Training Effects on Balance and Functional Performance Among Chronic Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Quds University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RESC/2023-11
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2023-06

CONDITIONS: Stroke; Chronic Stroke; Balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proactive balance training group (Active Comparator)
  Interventions: Other: proactive balance training
- Reactive balance training group (Active Comparator)
  Interventions: Other: Reactive balance training

INTERVENTIONS:
Other: proactive balance training — 20 participants will receive a proactive balance training program
  Arms: Proactive balance training group
Other: Reactive balance training — 20 participants will receive a Reactive balance training program
  Arms: Reactive balance training group

SUMMARY:
The study is an RCT study, comparing the proactive and reactive balance training among stroke survivors, the participants will be chronic stroke patients aged between 50- 75 years old, and the participants will receive a balance training program for 8 weeks 3 sessions in the week, the participants will randomly be allocated in two groups proactive group and the reactive group, at the end of the study will compare the different effects between proactive and reactive balance training

DETAILED DESCRIPTION:
The objectives of the study are: (1) To investigate the effect of reactive balance training on balance and functional performance, (2) To investigate the effect of proactive balance training on functional activity and balance stroke survivors, and (3) To study the reactive balance training versus the proactive balance on balance and functional performance among stroke survivors.

The study will be a single-blinded RCT study will consist of 40 chronic stroke patients and will allocate randomly into 2 groups, the first intervention group n=20 will have proactive-balance training, and the second group n= 20 will have reactive balance training, the two groups will be blinded.

The study population will be chronic stroke patients discharged from Bethlehem Arab Society for Rehabilitation (BASR), Alahli Hospital, Al Mezan Hospital, and Alehsan Society for Rehabilitation, and lives in Hebron City and their villages.

The program will consist of 24 sessions in 8 weeks, through 3 sessions weekly. The sessions will be 45 minutes, starting with a 10 Min warm-up exercise and then the balance training and the sessions will end with 5 Min cool-down exercise.

The session will be individualized, the program has sequences depending on the patient's ability.

The program consists of:

1. Sitting training
2. Standing training
3. Walking training The sequences of the training will be based on a balance training protocol.

ELIGIBILITY:
Inclusion Criteria:

1. chronic stroke patients
2. Males and females
3. Age from 50-75 years old
4. Able to follow up on instructions
5. Able to walk at least 10 meters continuously
6. Able to perform sub-maximal physical activity
7. stable health condition

Exclusion Criteria:

1. Acute stage or Subacute stage (less than 3 months)
2. stroke patients with other severe diseases
3. Head injuries
4. patients with mental problems
5. patients with vestibular problems
6. Patients refuse to sign the consent form

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire | 1 minute
  This measure assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in min-hours/week and time spent sitting. The short form consists of 7 questions, the questions ask about the time that patients spent being physically active in the last 7 days. The sequence of questions is from vigorous to moderate activities to walking then to sitting. And it is a valid and reliable questionnaire
Time Up and Go (TUG) | 1 minute
  Is a reliable and valid outcome measure.and it's a sensitive and specific test to measure balance and risk of fall among elderly. The patient will be sitting on chair with arm rest then will stand up and walk in straight line 3 m then will turns around and back to the chair and sit down, the timing will start when patient stand up from chair and ends when back to the chair and sit down.[33]
  The score of the TUG:
  1. ≤10s → completely independent
  2. ≤ 2s → Independent for main transfers
10 Meters walking test (MWT) | 5 minutes
  It is a reliable and vailed outcome measure, it is evaluated by measuring speed and counting the steps and time. The steps and time will be measured when patient start to walk from beginning point. Individual walks without assistance 10 meters (32.8 feet) and the time is measured for the intermediate 6 meters (19.7 feet) to allow for acceleration and deceleration.
The Falls Efficacy Scale (FES) | 2 minutes
  The FES was developed through a series of meetings between members of the Prevention of Falls. FES IS A confidence measure in performing a range of activities of daily living without falling. This scale has excellent reliability, is correlated with measures of balance and gait, and predicts future falls and decline in functional capacity. Most importantly, the FES has proven sensitive to change in fears following clinical interventions
Tinetti Balance Assessment tool or Tinetti Performance-Oriented Mobility Assessment (POMA) | 10 minutes
  It is a balancing tool with both a balance and a gait component that was created for the elderly. The balance component of the test evaluates the patient's ability to maintain postural control while standing, sitting statically, rising from a chair, immediately after standing, standing with eyes open and closed, turning 360 degrees, and during perturbation. The gait component evaluates the following during gait: symmetry, initiation, continuation, path, base of support, and postural sway. measures reactive balance by asking the patient to react to a perturbation.
  The test comprises 16 items:
  * 9 balance-related items and
  * 7 gait-related items
Mini-BESTest Balance Evaluation System Test (BEST) | 5 minutes
  The Mini-BESTest, the shorter version of the BESTest, was developed to reduce the assessment time. - 14-item Mini-BESTest is scored on a 3-level ordinal scale:
  * 0 : poor balance performance
  * 2: no balance impairment. Several studies have shown that the Mini-BESTest also was reliable and valid and useful for fall prediction. The use of the Mini-BESTest in community-dwelling people with chronic stroke has recently been reported, with excellent interrater and intrarater reliability and validity.
2 Minutes Walking test | 2 minutes
  There are 5 versions of walking tests available in the stroke population, the 12-, 6-, 5-, 3-, and 2-Minute Walk Tests.
  Will use 2 MWT:
  * To assess exercise tolerance in chronic airflow limitation.
  * Highly correlated with the 6 and 12 MWTs. A valid measure of self-selected walking speed.
  * The most time efficient.

CONTACTS AND LOCATIONS:
Locations (1):
- Amany, Hebron, West Bank, Palestinian Territories

IPD SHARING:
Plan to Share IPD: No